CLINICAL TRIAL: NCT03754387
Title: Mutil-institutions Comparing Antibiotic Therapy With Laparscopic Appendectomy in Pediatric Chronic Appendicitis
Brief Title: Antibiotic Therapy vs Laparscopic Appendectomy in Pediatric Chronic Appendicitis
Acronym: ATvsLAAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, zebing Zheng, Head of pediatric surgery, Zunyi Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZunyiMU
Record Dates: First submitted 2018-11-18; First posted 2018-11-27 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Chronic Appendicitis
Keywords: children; antibiotic therapy; laparoscopic appendectomy; randomized clinical trial(RCT); Chronic appendicitis
MeSH Terms: interventions — Ceftazidime; Appendectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic therapy group (Active Comparator): Ceftazidime will chosen as the antibiotic for this study because of its efficacy as a monotherapy for serious intraabdominal infections, requiring only a single, daily dose. Intravenous Ceftazidime sodium (50mg/kg/dose every 12 hours) is administered for 3 days to patients in the AT group, with the first dose given in the emergency department. The clinical status of patients in the AT group is reevaluated within 12 to 24 hours after admission by the surgeon on call. If the surgeon suspected progressive infection, perforated appendicitis, or peritonitis, the patient will underwent appendectomy. Intravenous antibiotic treatment will followed by 7 days of oral cefuroxime (250mg twice daily).
  Interventions: Drug: Ceftazidime
- Laparoscopic Appendectomy group (Experimental): Laparoscopic appendectomy will performed using. Prophylactic antibiotics (ceftazidime sodium 50mg/kg/dose ) will administered approximately 30 minutes before the incision was made. No further antibiotics will given to patients in the surgical group unless a wound infection was suspected postoperatively.
  Interventions: Procedure: appendectomy

INTERVENTIONS:
Drug: Ceftazidime — Patients choosing AT group were admitted to the hospital for observation and to receive intravenous antibiotics Intravenous Ceftazidime sodium (50mg/kg/dose every 12 hours) was administered for 3 days.
  Arms: Antibiotic therapy group
Procedure: appendectomy — APPT group consisted of admission to the hospital with promptinitiation of intravenous antibiotics and appendectomy
  Arms: Laparoscopic Appendectomy group

SUMMARY:
This clinical trial will compare antibiotic therapy with laparoscopic appendectomy in the treatment of pediatric chronic appendicitis in china. Enrolled patients will be randomised and an allocation ratio of 1:1 will be made via weighted minimisation, where half of the patients will receive antibiotic therapy with intravenous Ceftazidime sodium, while the other half will have a laparoscopic appendicectomy.

DETAILED DESCRIPTION:
In recent years, nonoperative treatment has challenged appendectomy as a first-line treatment of acute uncomplicated appendicitis by demonstrating its safety and short-term efficacy in adults. Several randomized controlled trials comparing appendectomy to antibiotics alone in children with acute uncomplicated appendicitis have been reported from other countries. These studies reveal that non-operative management of appendicitis is a safe treatment for appendicitis and is associated with a significantly lower risk of complications than appendectomy. However, the success rate of nonoperative management was 75% at 1year. Chronic appendicitis has been described as a possible cause of persistent right lower quadrant (RLQ) pain and laparoscopic appendectomy has been shown to benefit a large number of children，but there are no high-quality clinical trials. There are more than 200 million children in China. According to preliminary clinical data, the incidence of pediatric appendicitis in China is higher than Europe and America. Due to the Chinese parents have different cultures and educational backgrounds, more high-quality clinical trials are needed to guide parents to choose appropriate treatment for chronic appendicitis in children. Therefore, the investigators propose a multi-institutional trial in which patients and their families choose between antibiotics therapy (AT group) or laparoscopic appendectomy (LAAPT group) to chronic appendicitis in children aged 3-15 years. The investigators hypothesize that laparoscopic appendectomy will be successful in 90% of patients at 1 year follow-up and will be associated with fewer disability days, higher quality of life scores, and higher pain reduce scores than antibiotic therapy. This study will enroll 200 patients, age 3-15 years, with chronic appendicitis at 8-10 hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were eligible if they were between 3 and 15 years of age, and they suffered from chronic appendicitis.
2. US showing hyperemia and fecalith, ≤ 1.1 cm in diameter, compressible or non-compressible, no abscess, no phlegmon or CT showing hyperemia and fecalith, fat stranding, ≤ 1.1 cm in diameter, no abscess, no phlegmon.

Exclusion Criteria:

1. Exclusion criteria consisted of (a history of) chronic back pain
2. previous abdominal surgery (with the exception of diagnostic laparoscopies or a laparoscopic sterilization)
3. specific gastro-intestinal entities (such as inflammatory bowel disease) 4.gynaecological disease (all female patients consulted a gynaecologist)

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | 1 year
  The primary end point for patients in the antibiotic therapy group is resolution of chronic appendicitis, resulting in discharge from the hospital without the need for surgical intervention and no recurrent appendicitis during a minimum follow-up of 1 year (treatment efficacy). Treatment success in the laparoscopic appendectomy group is defined as a patient successfully undergoing an laparoscopic appendectomy and no recurrent abdominal pain during a minimum follow-up of 1 year (treatment efficacy).

SECONDARY OUTCOMES:
The rate of recurrence | 1 year
  late recurrence (after 1 year) of chronic appendicitis after conservative treatment, length of hospital stay and the amount of sick leave used by the patient.
postintervention pain scores | 1 year
  postintervention pain scores (VAS score range, 0-10; a score of 0 indicates no pain and 10 indicates the worst possible pain), and the use of pain medication.
Wound infection | 30 days
  Postintervention complications included clinical wound infection (surgical site infection) occurring within 30 days after the operative procedure as diagnosed by a surgeon or with a positive bacterial culture.
pneumonia | 7days
  Postintervention complication included pneumonia occurring within 7days after the operative procedure as diagnosed by clinical presentation and chest X-ray or CT-scan.
Diarrhea | 7 days
  Adverse effects of the antibiotic treatment during the conservation treatment
Incisional hernia | 1 year
  Postintervention complication included incisional hernia occurring within1year after the operative procedure as diagnosed by surgeon .
Bowel obstruction | 1 year
  Postintervention complication included bowel obstruction occurring within1year after the operative procedure as diagnosed by clinical presentation and abdominal X-ray or CT-scan.
persistent abdominal or incisional pain | 1 year
  Postintervention complication included persistent abdominal or incisional pain occurring within1year after the operative procedure as diagnosed by surgeon .

CONTACTS AND LOCATIONS:
Overall Officials: yuanmei Liu, Study Chair — Zunyi Medical College; peihong Yan, MD, Study Director — Children's hospital of guiyang; Shengli Gu, MD, Study Director — Zunyi First People's Hospital; Lei Geng, MD, Study Director — Affiliated hospital of Binzhou; Ziyong Li, MD, Study Director — Children's hospital of Dalian; Guoqing He, MD, Study Director — People's Hospital of Anshun City of Guizhou Province; Xuanzao Wu, MD, Study Director — Medical university of Guizhou; Guohong Yang, Study Director — people hospital of Suiyang
Locations (3):
- China (3):
  - children's hospital of Guiyang, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The first people hospital of zunyi, Zunyi, Guizhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minneci PC, Mahida JB, Lodwick DL, Sulkowski JP, Nacion KM, Cooper JN, Ambeba EJ, Moss RL, Deans KJ. Effectiveness of Patient Choice in Nonoperative vs Surgical Management of Pediatric Uncomplicated Acute Appendicitis. JAMA Surg. 2016 May 1;151(5):408-15. doi: 10.1001/jamasurg.2015.4534. PMID 26676711
- [Background] Anderson KT, Bartz-Kurycki M, Austin MT, Kawaguchi A, John SD, Kao LS, Tsao K. Approaching zero: Implications of a computed tomography reduction program for pediatric appendicitis evaluation. J Pediatr Surg. 2017 Dec;52(12):1909-1915. doi: 10.1016/j.jpedsurg.2017.08.050. Epub 2017 Sep 5. PMID 28927978
- [Background] Salminen P, Paajanen H, Rautio T, Nordstrom P, Aarnio M, Rantanen T, Tuominen R, Hurme S, Virtanen J, Mecklin JP, Sand J, Jartti A, Rinta-Kiikka I, Gronroos JM. Antibiotic Therapy vs Appendectomy for Treatment of Uncomplicated Acute Appendicitis: The APPAC Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2340-8. doi: 10.1001/jama.2015.6154. PMID 26080338